CLINICAL TRIAL: NCT03790254
Title: Oral D Mannose in the Prevention and Treatment of Recurrent Urinary Tract Infections: a Systematic Review
Brief Title: D Mannose for Prevention and Treatment of RUTIs
Acronym: mannoseRUTIs
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Daniele Porru, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: ReviewUTIs
Record Dates: First submitted 2018-12-26; First posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Recurrent Urinary Tract Infections; Antibiotic Prophylaxis; Antibiotic Resistance
Keywords: recurrent urinary tract infections; d mannose prophylaxis; antibiotic prophylaxis
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: systematic review

SUMMARY:
The aim of this review is to address clinical reliability, efficacy and safety of long-term treatment with oral D Mannose for the prevention of recurrent urinary tract infections (RUTIs) in females.

DETAILED DESCRIPTION:
A comprehensive systematic MEDLINE, Embase, Cochrane search was performed for English language reports published before December 2018 using the term "recurrent urinary tract infections and d mannose." We searched Medline, Embase, and the Cochrane Register of Controlled Trials since January 2010 to December 2018. Eligible studies did not include non-oral therapy, local (vaginal) treatment in women with RUTIs.

Study eligibility criteria- We identified eligible original articles. The heterogeneity of the available studies, their different rationale and aim, the assumption of d mannose for prophylaxis or treatment of recurrent UTIs need to be taken into account.

ELIGIBILITY:
Inclusion Criteria:

recurrent urinary tract infections (RUTIs)

Exclusion Criteria:

Upper urinary tract infections, severe clinical symptoms, fever > 37,5 with lumbar pain

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Search strategy and selection criteria Only publications with the text and/or the abstract written in the English language were considered. Additional papers cited in the references of the search manuscripts were further examined. Articles not addressing topics of interest were excluded, and the full text of the remaining articles was examined. Our literature search identified 15 articles pertaining to the search terms (Word variations have been searched). Further analysis of these articles resulted in 11 clinical trials which were deemed relevant to our review. The retrieved studies were assessed for their relevance based on the title and abstracts. Finally, studies references were screened in order to identify eventually unknown studies.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-25 (Actual)

PRIMARY OUTCOMES:
research literature data on d mannose for prevention and treatment of recurrent urinary tract infections. | January 2010-December 2018
  literature search of the Medline, Embase, and Cochrane Library databases

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Porru, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Urology Department Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No